CLINICAL TRIAL: NCT04920942
Title: Ivermectin Treatment Efficacy in Covid-19 High Risk Patients (I-TECH Study): A Multicenter Open-label Randomized Controlled Trial
Brief Title: Ivermectin Treatment Efficacy in Covid-19 High Risk Patients
Acronym: I-TECH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clinical Research Centre, Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I-TECH21
Record Dates: First submitted 2021-05-31; First posted 2021-06-10 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
Keywords: Ivermectin; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-label, randomized controlled clinical trial involving COVID-19 designated hospitals in Malaysia. Patients are randomized at ratio of 1:1 to groups receiving ivermectin for 5 days plus standard-of-care versus standard-of-care only. Patients will be assigned to stratified randomized treatments based on a central, computer-generated randomization scheme coordinated by an independent third party. Based on national guidelines, all high risk COVID-19 patients will be admitted to hospitals, and allow discharge once criteria met
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Ivermectin 0.4mg/kg/day for 5 days + standard-of-care
  Interventions: Drug: Ivermectin 0.4mg/kg/day for 5 days
- Control group (No Intervention): Standard-of-care only

INTERVENTIONS:
Drug: Ivermectin 0.4mg/kg/day for 5 days — Ivermectin 0.4mg/kg/day for 5 days with standard-of-care
  Arms: Treatment group

SUMMARY:
This is a multicenter study, which is aimed to investigate the efficacy of the Ivermectin drug in high risk COVID-19 patients. This study will compare Ivermectin treatment efficacy with standard of care alone. Target cohort is mild to moderate symptomatic Covid-19 (Stage 2-3), high risk patients aged 50 years and above with comorbidity, who presented to hospitals within first 7 days of illness.

DETAILED DESCRIPTION:
Objectives

Primary Objective:

To assess the effectiveness of Ivermectin in preventing progression of Covid-19 to severe disease (clinical stage 4 or 5), which is defined as severe pneumonia requiring oxygen supplement or critically ill requiring intensive care.

Secondary Objectives:

1. To assess the efficacy of Ivermectin in reducing mortality rate among high risk COVID-19 patients.
2. To compare difference in resolution of symptoms, chest radiograph, laboratory investigations, ICU admission, mechanical ventilation and length of hospital stay.

Methodology Study Type and Design This is a multicenter, open-label, randomized controlled clinical trial involving COVID-19 designated hospitals in Malaysia. Patients are randomized at ratio of 1:1 to groups receiving ivermectin for 5 days plus standard-of-care versus standard-of-care only. Patients will be assigned to stratified randomized treatments based on a central, computer-generated randomization scheme coordinated by an independent third party. Based on national guidelines, all high risk COVID-19 patients will be admitted to hospitals, and allow discharge once criteria are met.

Rationale of ivermectin dose and duration in this study:

The dose regimens used in various randomized control trials with positive results range from 0.2mg/kg single dose to 0.6mg/kg/day for 5 days 10-15. PK/PD studies have shown that the antiviral effect of Ivermectin is dose dependent 9,15. As SARS-CoV-2 viral load peaks during the first week of illness and may prolong in severe disease 18, we believe a high dose of ivermectin 0.4mg/kg/day for 5 days would be reasonable and safe to achieve our study objectives.

Standard of care:

Based on the current Malaysian guidelines, standard of care for mild to moderate Covid-19 patients includes isolation, infection control, close monitoring (clinical findings, laboratory tests, chest imaging) and symptomatic treatment.

Study Population The population for this clinical trial will be comprised of adults with a polymerase chain reaction (PCR) confirmed diagnosis of COVID-19 admitted to any of the participating hospitals. Participants who

1. Treatment group: Ivermectin 0.4mg/kg/day for 5 days + standard-of-care
2. Control group: Standard-of-care only

Patients who fulfil the inclusion criteria and do not meet the exclusion criteria will be enrolled. Identification of eligible participants will be done prospectively at each study site.

Sample Size Sample size calculation was performed using ScalexProp Version 1.0.2 (Naing, 2016). The calculation is based on superiority trial design and the primary outcome measure of the need to have supplemental oxygen therapy during the hospital admission. We regard a 9% difference between intervention arm and control arm as a clinically important outcome. Based on local data, 17.5% of COVID-19 aged 50 years and above, with stage 2 and 3 disease and comorbidity, progressed to severe disease 3. The need of supplemental oxygen therapy is expected to be about 8.8% in intervention arm and 17.5% in control arm. With a margin of superiority set to be 1%, the study requires 231 patients for each arm or in total 462 patients. Considering potential dropouts during the trial, we would require up to 500 patients or 250 patients each arm. The sample size provides a level of significance at 5% with 80% power (2-sided test).

ELIGIBILITY:
Inclusion Criteria:

1. RT-PCR or antigen test confirmed COVID-19 cases
2. Aged 50 years and above,with at least one co-morbidities*
3. Within the first 7 days of illness (from symptom onset)
4. Mild to moderate clinical severity

Exclusion Criteria:

1. Asymptomatic stage 1 patients
2. Patients with SpO2 less than 95% at rest. (unless it is an expected baseline SpO2 due to preexisting disease, eg. COAD or pulmonary fibrosis)
3. Patients who need oxygen supplements
4. Patients with concomitant bacterial, fungal, parasitic or other viral infections prior to enrollment.
5. Patients with severe hepatic impairment (>Grade 3: ALT >10 times of upper normal limit)
6. Malabsorptionsyndromeorotherclinicallysignificantgastrointestinaldisease that may affect absorption of the study drug (non-correctable vomiting, diarrhea, ulcerative colitis, and others).
7. Pregnant or nursing women.
8. Female patients of reproductive age who cannot consent to contraceptive use of oral contraceptives, mechanical contraceptives such as intrauterine devices or barrier devices (pessaries, condoms), or a combination of these devices from the start of ivermectin administration to 7 days after the end of ivermectin administration.
9. Male patient who has female partner of reproductive age and he cannot agree to use contraception from the start of ivermectin treatment till 7 days after treatment.
10. Patients receiving chemotherapy
11. Patients who received interferon or drugs with reported antiviral activity against COVID-19 (favipiravir, hydroxychloroquine sulfate, chloroquine phosphate, lopinavir-ritonavir combination, remdesivir) in the past 7 days before enrollment.
12. Patients in whom this episode of infection is a recurrence or reinfection of COVID- 19.
13. Patients who have previously received ivermectin.
14. Patient receiving warfarin or any medications known to interact with ivermectin.
15. Acute medical or surgical emergency (eg. DKA/MI/stroke).
16. Other patients judged ineligible by the principal investigator or sub-investigator.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Patients who Progressed to Severe Disease (Clinical stage 4 or 5) | Within 28 days since administered Ivermectin
  The number of patients recruited who clinically deteriorated to clinical stage 4 or 5. The differences between two study arms will be assessed via chi-square test. Estimates will be reported in proportions and 95% confidence intervals, together with their corresponding p-values. A logistic regression will also be performed, to enable estimates to be presented in the form of odds ratio and its corresponding 95% confidence interval, potentially adjusting for clinically relevant and statistically significant variable
Time Required for Patients on Treatment Arm to Progressed to Severe Disease (Clinical stage 4 or 5) | Within 28 days since administered Ivermectin
  The time duration for patients in the treatment arm to deteriorated to clinical stage 4 or 5. The differences between two study arms will be assessed via chi-square test. Estimates will be reported in proportions and 95% confidence intervals, together with their corresponding p-values. A logistic regression will also be performed, to enable estimates to be presented in the form of odds ratio and its corresponding 95% confidence interval, potentially adjusting for clinically relevant and statistically significant variable

SECONDARY OUTCOMES:
Mortality | Through study completion, an average of 28 days
  The number of died patients were evaluated in study and control groups. The differences between two study arms will be assessed via chi-square test. Estimates will be reported in proportions and 95% confidence intervals, together with their corresponding p-values. A logistic regression will also be performed, to enable estimates to be presented in the form of odds ratio and its corresponding 95% confidence interval, potentially adjusting for clinically relevant and statistically significant variable
Number of Participants with Complete Resolution of Symptoms by day 5 of Enrolment | 5 days since time of recruitment
  The total numbers of patients with complete resolution of symptoms were evaluated in study and control groups. The differences between two study arms will be assessed via chi-square test. Estimates will be reported in proportions and 95% confidence intervals, together with their corresponding p-values. A logistic regression will also be performed, to enable estimates to be presented in the form of odds ratio and its corresponding 95% confidence interval, potentially adjusting for clinically relevant and statistically significant variable
Chest Radiograph Changes Pertaining to COVID-19 by Day 5 of Enrolment | 5 days since time of recruitment
  Radiological Changes Pertaining to COVID-19 is recorded at day 1 of enrolment and compared with day 5 of enrolment. The differences between two study arms will be assessed via chi-square test. Estimates will be reported in proportions and 95% confidence intervals, together with their corresponding p-values. A logistic regression will also be performed, to enable estimates to be presented in the form of odds ratio and its corresponding 95% confidence interval, potentially adjusting for clinically relevant and statistically significant variable
Changes in Serum Absolute Lymphocyte Count | From starting to the end of ivermectin therapy (0 to end of 5th day)
  For changes in Serum Absolute Lymphocyte counts (cell/mm3), baseline values, value at each post baseline analysis, changes from baseline at each post baseline analysis will be provided descriptively by each study arm either in mean and SD or median and interquartile range.
Changes in Serum Absolute Neutrophil Counts | From starting to the end of ivermectin therapy (0 to end of 5th day)
  For changes in Serum Absolute Neutrophil counts (cell/mm3), baseline values, value at each post baseline analysis, changes from baseline at each post baseline analysis will be provided descriptively by each study arm either in mean and SD or median and interquartile range.
Changes in Serum C-Reative Protein (CRP) | From starting to the end of ivermectin therapy (0 to end of 5th day)
  For changes in Serum C-Reative Protein (mg/L), baseline values, value at each post baseline analysis, changes from baseline at each post baseline analysis will be provided descriptively by each study arm either in mean and SD or median and interquartile range.
Changes in Serum Creatinine | From starting to the end of ivermectin therapy (0 to end of 5th day)
  For changes in Serum Creatinine (micro mol/L), baseline values, value at each post baseline analysis, changes from baseline at each post baseline analysis will be provided descriptively by each study arm either in mean and SD or median and interquartile range.
Changes in Serum Alanine Aminotransferase (ALT) | From starting to the end of ivermectin therapy (0 to end of 5th day)
  For changes in Serum Alanine Aminotransferase (U/L), baseline values, value at each post baseline analysis, changes from baseline at each post baseline analysis will be provided descriptively by each study arm either in mean and SD or median and interquartile range.
Numbers of Participants Admitted to the Intensive Care Unit | Through study completion, an average of 28 days
  The number of patients admitted to the intensive care unit were evaluated in study and control groups
Numbers of Participants who Require Mechanical Ventilation | Through study completion, an average of 28 days
  The number of patients who require mechanical ventilation were evaluated in study and control groups
The Length of Hospital Stay (in Calendar days) | Through study completion, an average of 28 days
  The average number of hospitalisation required for both groups.
Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | From the 6th day of study to the 28th day of study
  Adverse effects of ivermectin

CONTACTS AND LOCATIONS:
Overall Officials: CHEE L LIM, MRCP, Principal Investigator — Ministry of Health, Malaysia
Locations (21):
- Malaysia (21):
  - Sultanah Aminah Hospital, Johor Bahru, Johor
  - Sultanah Bahiyah Hospital, Alor Star, Kadah
  - Sultan Abdul Halim Hospital, Sungai Petani, Kedah
  - Hospital Raja Permaisuri Bainun, Ipoh, Ipoh, Perak
  - Taiping Hospital, Taiping, Perak
  - Tuanku Fauziah Hospital, Kangar, Perlis
  - Pulau Pinang Hospital, George Town, Pulau Pinang
  - Lahad Datu Hospital, Tawau, Sabah
  - Sarawak General Hospital, Kuching, Sarawak
  - Sungai Buloh Hospital, Shah Alam, Selangor
  - Permai Hospital, Kempas
  - Kepala Batas Hospital, Kepala Batas
  - Kuala Kangsar Hospital, Kuala Kangsar
  - Kuala Lumpur Hospital, Kuala Lumpur
  - Sultanah Nur Zahirah, Kuala Terengganu
  - Melaka Hospital, Malacca
  - Putrajaya Hospital, Putrajaya
  - Duchess of Kent Hospital, Sandakan
  - Low Risk COVID-19 Quarantine & Treatment Centre - Malaysia Agro Exposition Park Serdang (MAEPS), Serdang
  - Sg Siput Hospital, Sungai Siput
  - Tumpat Hospital, Tumpat

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim SCL, Hor CP, Tay KH, Mat Jelani A, Tan WH, Ker HB, Chow TS, Zaid M, Cheah WK, Lim HH, Khalid KE, Cheng JT, Mohd Unit H, An N, Nasruddin AB, Low LL, Khoo SWR, Loh JH, Zaidan NZ, Ab Wahab S, Song LH, Koh HM, King TL, Lai NM, Chidambaram SK, Peariasamy KM; I-TECH Study Group. Efficacy of Ivermectin Treatment on Disease Progression Among Adults With Mild to Moderate COVID-19 and Comorbidities: The I-TECH Randomized Clinical Trial. JAMA Intern Med. 2022 Apr 1;182(4):426-435. doi: 10.1001/jamainternmed.2022.0189. PMID 35179551